CLINICAL TRIAL: NCT04840212
Title: The Effectiveness of Aromatherapy in an Urban, Safety-Net Hospital on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Justin Buchert, Quality Specialist, Parkland Health and Hospital System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU-2020-1176
Record Dates: First submitted 2021-03-24; First posted 2021-04-09 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Patients currently hospitalized in multiple service lines (surgical intensive care unite [SICU], surgical progressive care unit [SPCU], burns, trauma, plastics, general surgery, orthopedics, surgical specialties, and inpatient rehabilitation) will be included. Lavender-Sandalwood scented aromatherapy sticker will be used throughout the patient hospital stay.
  Interventions: Other: Lavender-Sandalwood scented aromatherapy sticker
- Control Group (No Intervention): The historical control group will be comprised of hospitalized patients in multiple service lines from the previous year with the same time period, demographic characteristics, service line, and relevant clinical information.

INTERVENTIONS:
Other: Lavender-Sandalwood scented aromatherapy sticker — The Lavender-Sandalwood scented aromatherapy sticker will be placed on the patient gown.
  Arms: Study Group

SUMMARY:
The purpose of this project is to evaluate the effectiveness of aromatherapy on reducing pain in the acute care setting at Parkland Health and Hospital System. The target population for this study will be patients who are recovering from surgical procedures and are in the Surgical Services inpatient units.

DETAILED DESCRIPTION:
This study will evaluate the impact of aromatherapy on the administration of opioid pain medication administration among the inpatient Surgical Services population. Patients from multiple units (burns, trauma, plastics, general surgery, and orthopedics) will be included. The study duration will be six months.

The Lavender-Sandalwood scented aromatherapy sticker has been selected for this study because it helps promote relaxation, comfort, and sleep. After introducing the patient to the study and obtaining informed consent for participation, the sticker will be placed on the patient gown. The sticker aroma last for twelve (12) hours and can be replaced upon patient request. The sticker will be used for 72 hours after the surgical procedure and initiated during patient's hospital stay. After use of aromatherapy sticker, the patient will participate in a survey to evaluate their experience with the sticker. In addition, opioid pain medication administration will be collected along with demographic and relevant clinical information.

The historical control group will be comprised of hospitalized patients from the previous year with the dame time period, demographic characteristics, service line, and relevant clinical information. Other methods for establishing a control group (a randomized controlled trial or concurrent case control study) are not feasible due to the potential impact of the aromatherapy on all patients in close proximity to the enrolled patient. The historical control cohort will also allow to collect non-COVID time period data to avoid any bias due to the pandemic.

The primary endpoint for this study is a decrease in the percentage of study patients who are in the pain scale threshold from 7-10 requiring opioid pain medication administration 72 hours after surgery/intervention. The pain score will be recorded for each patient before opioid pain medication administration within the time period. The historical control group will be from the same precious year time frame to control for any seasonal bias. The first dose or baseline pain score will be collected for each group and other relevant pain scores within the 72-hour time period after surgery. Demographic and other clinically relevant information will be compared between study and historical control group to account for any differences in the primary and secondary outcomes.

Outcomes will be collected from the electronic medical record (pain scores, opioid pain medication administration, and length of stay by service line. Qualitative measures of aromatherapy effectiveness will be obtained through patient surveys.

Data to be extracted for the active current group and the historical matched control group include the following:

* Patient demographics (matching variable list)

  * Age (18-29, 30-39, 40-49, 50-59, 60-69, >70.
  * Gender
  * Race/ethnicity
* Other demographic variables not proposed in matching

  * Diabetes
  * High blood pressure
  * Other clinical co-morbidities
* Clinical history

  * Opioid pain medication administration given for 72 hours after surgery or intervention
  * Surgical Service Units: burns, trauma, plastics, general surgery, orthopedics
  * Dates of admission and discharge
  * Length of stay
  * Date and type of surgery/intervention
  * All Pain scores within 72 hours after surgery or intervention.

Data to be extracted for the current active group:

* Dates of aromatherapy application (possible 6 doses within 72-hour time period)
* Patient survey forms

ELIGIBILITY:
Inclusion Criteria:

A) For the current study group:

* Inpatients, 18 years and older, admitted to a surgical service inpatient unit and who are experiencing pain and/or anxiety, and
* No history of chronic pain, respiratory problems, asthmas, allergies, or lost sense of smell, and
* Provide informed consent to participate in the study, and
* Complain of pain and anxiety in the 72 hours after surgery or intervention and requiring PANX.

B) For the historical control group:

• Patients from the same time in the previous year with the same inclusion and exclusion criteria.

Exclusion Criteria:

A) For the current study group:

* Patients with known allergies or sensitivities to aromatherapy products.
* Lack of interest in participating in or subsequent withdrawal from the research.
* Patients who are intubated, have died, or had serious disease complications will also be excluded from the study time period and previous year historical control group.

Subject withdrawal from the Study

* Patients who develop allergic symptoms while the aromatherapy patch is applied.
* Patients who require intubation or critical interventions during their hospitalization.

B) For the historical control group:

• Anyone who does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Number of participants who needed opioid pain medication administration after surgery | 72 hours after surgery
  Pain scale is measured by patients verbal report of pain and ranges from 0 to 10 , with higher scores indicating more pain and thus a worse outcome.

SECONDARY OUTCOMES:
Mean duration of hospital stay | 6 months
  Duration of hospital stay will be collected from the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Buchert, MSN, M.Ed., MS, RN, Principal Investigator — Parkland Health and Hospital System
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No